CLINICAL TRIAL: NCT03481647
Title: Evaluation of an Oral Care Programme for Patients Undergoing Treatment for Head and Neck Cancer Regarding Mucositis, Oral Health, Epigenetic Modifications, Patient-related Factors, Quality of Life and Health Economy
Brief Title: Evaluation of an Oral Care Programme for Head and Neck Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Ryhov County Hospital (Other); Region Jönköping County (Other Government); Swedish Cancer Foundation (Other); Kalmar County Hospital (Other); Norrlands University Hospital (Other); The Sjöberg Foundation (Unknown); TUA research funding: The Sahlgrenska Academy/Region Västra Götaland (Unknown); Malmö University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 831-16
Record Dates: First submitted 2018-01-16; First posted 2018-03-29 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention group: intensified oral care programme Control group: conventional oral care
Who Masked: Participant
Masking Description: The participants will not be aware of the care/treatment given to the other group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The intervention consists of professional oral care and swabbing of the mucosal membranes with a saline and bicarbonate solution, five daily rinses with a saline and bicarbonate solution, a diary to register oral care measures and rinses
  Interventions: Procedure: Oral care programme
- Control (No Intervention): Professional oral care once a week according to existing routine

INTERVENTIONS:
Procedure: Oral care programme — Professional oral care (dental hygienist), intensified oral care measures by the patient
  Arms: Intervention

SUMMARY:
This study will evaluate the effect of an intensified oral care programme on prevalence, severity and duration of mucositis in patients undergoing treatment for cancer in the head and neck region.

Patients in the control group get professional oral care once a week.

DETAILED DESCRIPTION:
This study will evaluate the effect of an oral care programme on prevalence, severity and duration of mucositis in patients undergoing treatment for cancer in the head and neck region. The oral care programme consists of professional oral care and swabbing of the mucosal membranes with a saline/bicarbonate solution once a week. The patients are instructed to rinse with a saline/bicarbonate solution 5 times per day. They are given an oral care diary to help them keep track of their daily oral hygiene measures and rinses. Repeated oral hygiene instructions are given if needed.

Patients in the control group get professional oral care once a week.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to receive full dose of curative RT including major salivary glands in the radiation field

Exclusion Criteria:

* Patients with recurrent cancer
* Patients with severe cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral mucositis | First week of RT (mucositis score at one time-point)
  Reduced incidence of clinical mucositis assessed using Oral Mucositis Assessment Scale (9 areas in the mouth are examined and signs of ulceration are scored; 0=no lesion,1= lesion <1cm2, 2=lesion 1-3 cm2, 3=lesion > 3 cm2 as well as erythema, which is scored as follows: 0=no erythema, 1= mild erythema and 2=severe erythema. Total score for ulceration can vary from 0-27 and for erythema from 0-18. Mucositis is present at scores ≥ 1.)
Oral mucositis | Second week of RT (mucositis score at one time-point)
  Reduced incidence of clinical mucositis assessed using Oral Mucositis Assessment Scale (9 areas in the mouth are examined and signs of ulceration are scored; 0=no lesion,1= lesion <1cm2, 2=lesion 1-3 cm2, 3=lesion > 3 cm2 as well as erythema, which is scored as follows: 0=no erythema, 1= mild erythema and 2=severe erythema. Total score for ulceration can vary from 0-27 and for erythema from 0-18. Mucositis is present at scores ≥ 1.)
Oral mucositis | Third week of RT (mucositis score at one time-point)
  Reduced incidence of clinical mucositis assessed using Oral Mucositis Assessment Scale (9 areas in the mouth are examined and signs of ulceration are scored; 0=no lesion,1= lesion <1cm2, 2=lesion 1-3 cm2, 3=lesion > 3 cm2 as well as erythema, which is scored as follows: 0=no erythema, 1= mild erythema and 2=severe erythema. Total score for ulceration can vary from 0-27 and for erythema from 0-18. Mucositis is present at scores ≥ 1.)
Oral mucositis | Fourth week of RT (mucositis score at one time-point)
  Reduced incidence of clinical mucositis assessed using Oral Mucositis Assessment Scale (9 areas in the mouth are examined and signs of ulceration are scored; 0=no lesion,1= lesion <1cm2, 2=lesion 1-3 cm2, 3=lesion > 3 cm2 as well as erythema, which is scored as follows: 0=no erythema, 1= mild erythema and 2=severe erythema. Total score for ulceration can vary from 0-27 and for erythema from 0-18. Mucositis is present at scores ≥ 1.)
Oral mucositis | Fifth week of RT (mucositis score at one time-point)
  Reduced incidence of clinical mucositis assessed using Oral Mucositis Assessment Scale (9 areas in the mouth are examined and signs of ulceration are scored; 0=no lesion,1= lesion <1cm2, 2=lesion 1-3 cm2, 3=lesion > 3 cm2 as well as erythema, which is scored as follows: 0=no erythema, 1= mild erythema and 2=severe erythema. Total score for ulceration can vary from 0-27 and for erythema from 0-18. Mucositis is present at scores ≥ 1.)
Oral mucositis | Sixth week of RT (mucositis score at one time-point)
  Reduced incidence of clinical mucositis assessed using Oral Mucositis Assessment Scale (9 areas in the mouth are examined and signs of ulceration are scored; 0=no lesion,1= lesion <1cm2, 2=lesion 1-3 cm2, 3=lesion > 3 cm2 as well as erythema, which is scored as follows: 0=no erythema, 1= mild erythema and 2=severe erythema. Total score for ulceration can vary from 0-27 and for erythema from 0-18. Mucositis is present at scores ≥ 1.)

CONTACTS AND LOCATIONS:
Overall Officials: Annica Almståhl, Assoc.prof, Principal Investigator — Göteborg University
Locations (2):
- Sweden (2):
  - Institute of odontology, Gothenburg
  - Länssjukhuset Ryhov, Jönköping

IPD SHARING:
Plan to Share IPD: No
We are not planning to make IPD available to researchers not involved in the project